CLINICAL TRIAL: NCT06198712
Title: A Single Arm, Open Label, Phase 1/2 Study to Evaluate the Pharmacokinetics and Safety of Etavopivat in Pediatric Patients With Sickle Cell Disease
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of Etavopivat in Pediatric Patients With Sickle Cell Disease
Acronym: HIBISCUS KIDS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Forma Therapeutics, Inc. (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4202-HEM-202; 2022-001689-36 (EudraCT Number)
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Etavopivat (Experimental): Participants will receive Etavopivat once daily (QD) orally.
  Interventions: Drug: Etavopivat

INTERVENTIONS:
Drug: Etavopivat — Participants will receive oral tablets of etavopivat once daily.

SUMMARY:
This study is being done to learn about etavopivat, a once a day medicine taken by mouth in adolescents with sickle cell disease. The main goals are to study safety and how long etavopivat stays in the bloodstream, while also studying if there are benefits from taking etavopivat. Eligible participants who enter the study will start a 96-week treatment period. At the end of the 96 weeks, participants will have an end of study visit that occurs 4 weeks later. The participants will receive etavopivat every day throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Type of Participant and Disease Characteristics

  1. Patient has confirmed diagnosis of SCD

     • Documentation of SCD genotype (HbSS, HbSβ0-thalassemia or other sickle cell syndrome variants) based on prior history of laboratory testing. Molecular genotyping is not required. SCD genotype may be determined from the results of Hb electrophoresis, high-performance liquid chromatography (HPLC), or similar testing. Note that Hb electrophoresis is performed by the local laboratory at Screening.
  2. Hemoglobin greater than or equal to (≥) 5.5 and less than (<) 10.5 grams per deciliter (g/dL)
  3. Adolescent patients with severe SCD, as defined by at least 1 of the following:

     * Two or more VOCs in the past 12 months, defined as a previously documented episode of acute chest syndrome (ACS) or acute painful crisis (for which there was no explanation other than VOC) which required prescription or healthcare professional-instructed use of analgesics for moderate to severe pain
     * Hospitalization for any SCD-related complication in the last 12 months
     * Proteinuria, defined as an albumin:creatinine ratio (ACR) > 100 milligrams per gram (mg/g) on 2 measures (separated by ≥ 1 month) as an indicator of early renal disease
     * History of a conditional TCD in the last 12 months, but not currently being treated with chronic transfusion therapy. Conditional TCD is defined as a TAMMV of 170-199 centimeters per second (cm/s) by TCD or 155-184 cm/s by imaging TCD (TCDi).
  4. For participants taking hydroxyurea (HU), the dose of HU (mg/kg) must be stable (no more than a 20% change in dosing) for at least 90 days prior to start of study treatment with no anticipated need for dose adjustments during the study, in the opinion of the Investigator
  5. Patients on crizanlizumab or L-glutamine treatment at the time of consent may be eligible if they:

     * Have been on a stable dose for ≥ 12 months at the time of consent (ie, no changes to the dose except for changes to weight or for safety reasons)
     * For patients on crizanlizumab, have been ≥ 80% compliant with the planned regimen during the 12 months prior to the time of consent

Exclusion Criteria:

* Medical Conditions

  1. More than 10 VOCs within the past 12 months that required a hospital, emergency room (ER), or clinic visit
  2. Hospitalized for sickle cell crisis or other vaso-occlusive event within 14 days of Screening
  3. Abnormal TCD in the prior 12 months

     Prior/Concomitant Therapy
  4. Patients receiving regularly scheduled blood (RBC) transfusion therapy (also termed chronic, prophylactic, or preventive transfusion)
  5. Received any blood products within 30 days of starting study treatment
  6. Receiving or use of concomitant medications that are strong inducers of cytochrome P450 (CYP) 3A4/5 within 2 weeks of starting study treatment
  7. Use of voxelotor within 28 days prior to starting study treatment or anticipated need for this agent during the study
  8. Receipt of erythropoietin or other hematopoietic growth factor treatment within 28 days of starting study treatment or anticipated need for such agents during the study
  9. Receipt of prior cellular based therapy (eg, hematopoietic cell transplant, gene modification therapy)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2028-02-23 (Estimated); Study Completion 2029-08-08 (Estimated)

PRIMARY OUTCOMES:
Single-dose: maximum plasma concentration (Cmax) | During the 24-week primary treatment period
Single-dose: area under the plasma concentration time curve from dosing (time 0) to time t ((AUC)0-t) | During the 24-week primary treatment period
Single-dose: area under the plasma concentration time curve from zero to time infinity (AUC0-inf) | During the 24-week primary treatment period
Steady-state maximum plasma concentration (Cmax,ss) | During the 24-week primary treatment period
Steady-state area under the concentration time curve over the dosing interval (AUCtau,ss) | During the 24-week primary treatment period
Steady-state average plasma concentration (Cavg,ss) | During the 24-week primary treatment period
Steady-state minimum plasma concentration (Cmin,ss) | During the 24-week primary treatment period
Incidence of adverse events (AEs), serious adverse events (SAEs), and AEs related to etavopivat | During the 24-week primary treatment period
Number of premature discontinuations | During the 24-week primary treatment period
Number of dose interruptions | During the 24-week primary treatment period
Number of dose reductions | During the 24-week primary treatment period

SECONDARY OUTCOMES:
Incidence of AEs, SAEs, and AEs related to etavopivat | During the 72-week treatment extension period
Number of premature discontinuations | During the 72-week treatment extension period
Number of dose interruptions | During the 72-week treatment extension period
Number of dose reductions | During the 72-week treatment extension period
Hemoglobin (Hb) response rate | Baseline, week 12 and 24
Change in Hb from baseline | Baseline, week 12 and 24
Change from baseline in number of vaso-occlusive crises (VOCs) | Baseline and week 24
Change from baseline in Annualized Rate of VOC | Baseline and week 24
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale | Baseline, week 12 and 24
  PROMIS is a 10-item patient-reported health outcome measurement system used to evaluate quality of life in both children and adults. The assessment is based on the responses - 1. Never, 2. Almost never, 3. Sometimes, 4. Often and 5. Almost always. 'Never' response on the PROMIS fatigue scale indicates better quality of life.
Change from baseline in time-averaged mean of the maximum velocity (TAMMV) by transcranial Doppler ultrasonography (TCD) | Baseline, week 24, 48, and 96

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (16):
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Hôpital Robert Debrè - APHP, Paris, France
- Kenya (4):
  - KEMRI-Walter-Reed Kericho, Kericho
  - Ahero Clinical Trials Unit, Kisumu, Kenya, Kisumu
  - Kombewa Clinical Research Centre, Kisumu
  - Kenya Medical Research Institute-Centre for Respiratory Disease Research, Siaya Clinical Research Annexe, Siaya
- Lebanon (2):
  - American University of Beirut Medical center, Beirut
  - Hospital Nini, Tripoli
- Nigeria (3):
  - University of Nigeria Teaching Hospital, Enugu, Enugu
  - Lagos University Teaching Hospital, Lagos, Lagos
  - Aminu Kano Teaching Hospital (AKTH), Tarauni
- Turkey (Türkiye) (2):
  - Hacettepe University pediatric hematology, Ankara
  - Acıbadem Adana Hastanesi, Seyhan
- United Kingdom (3):
  - Guys and St Thomas NHS Foundation Trust / Evelina Childrens Hospital, London
  - Kings College Hospital - Alex Mowat Research Hub, London
  - Manchester Royal Infirmary_1, Manchester

IPD SHARING:
Plan to Share IPD: Yes